CLINICAL TRIAL: NCT00336531
Title: Clinical Study to Evaluate the Efficacy of Prophylactic Itraconazole in High-Dose Chemotherapy and Autologous Hematopoietic Stem Cell Transplantation for Pediatric Solid Tumors
Brief Title: Efficacy of Prophylactic Itraconazole in High-Dose Chemotherapy and Autologous Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Ki Woong Sung, Samsng Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2006-02-069
Record Dates: First submitted 2006-06-11; First posted 2006-06-13 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Neuroblastoma; Brain Tumor; Retinoblastoma; Wilms Tumor; Mycoses
Keywords: prophylactic itraconazole; Relapsed pediatric solid tumors; Embryonal brain tumor
MeSH Terms: conditions — Neuroblastoma; Brain Neoplasms; Retinoblastoma; Wilms Tumor; Mycoses | interventions — Itraconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: itraconazole — 2.5 mg/kg twice daily for the first two days --> once daily

SUMMARY:
The purpose of this study is to investigate whether the prophylactic use of itraconazole is a better option than empirical use of itraconazole in the management (prevention and treatment) of fungal infection associated with high-dose chemotherapy and autologous hematopoietic stem cell transplantation in children with high-risk solid tumor.

DETAILED DESCRIPTION:
With the advance of chemoradiotherapy, survival of patients, especially children, with malignant disease has improved. However, prognosis is still poor with conventional chemotherapy if patients have an advanced or high-risk tumor at diagnosis. Outcome in advanced or high-risk pediatric solid tumor such as advanced neuroblastoma, high-risk brain tumor, or recurrent pediatric solid tumor is still not satisfactory with conventional chemotherapy. In this context, investigators have explored the possible efficacy of high-dose chemotherapy (HDCT) and autologous stem cell transplantation (ASCT) in patients with high-risk or relapsed pediatric solid tumor. Efficacy of HDCT and ASCT has been well demonstrated in high-risk neuroblastoma, high-risk brain tumor, and recurrent pediatric solid tumors. Therefore, now, HSCT and ASCT is the most important treatment modality in the treatment of a variety of pediatric solid tumors poorly responding to conventional chemotherapy.

However, although HDCT and ASCT has improved the survival of patients with high-risk tumor, a variety of clinical issues associated with HDCT and ASCT are present causing significant morbidity and even mortality. The most frequent cause of morbidity associated with HDCT and ASCT is infection. Once high-dose myeloablative chemotherapeutic agents are administered, most hematopoietic cells in bone marrow die and prolonged marrow aplasia is unavoidable even after autologous hematopoietic stem cells infusion because it takes time for infused stem cells to reconstitute sufficient hematopoietic function. In addition, high-dose chemotherapy results in severe gastrointestinal mucosal damage which facilitates bacterial and/or fungal infection via damaged mucosal barrier. Therefore, infection is a major cause of morbidity and mortality associated with HDCT and ASCT. Common pathogens associated with infection during HDCT and ASCT are bacteria and fungi.

To reduce the chance of infection and therefore, to reduce the morbidity and mortality from severe infection, various prophylactic antibiotics including antibacterial, antifungal, and antiviral agents have been used according to standard guideline in allogeneic stem cell transplantation. However, in autologous transplantation for solid tumor in which hematologic recovery is rapid and immune suppression is less severe than allogeneic transplantation, there is no standard guideline for the use of prophylactic antibiotics whereas infection is the most important cause of morbidity. Standard guideline for the use of prophylactic antifungal agent is also not available. While some institutes use anti-fungal agent prophylactically, others use antifungal agent empirically only when neutropenic fever persist despite of empirical use of antibacterial agents.

HDCT in pediatric solid tumor is generally more intensive, and therefore, usually cause more severe mucositis than that in adult tumor. Severe mucositis facilitates fungal infection via damaged mucosal barrier (mainly by Candida species). Therefore, use of prophylactic anti-fungal agent may reduce the morbidity and mortality associated with HDCT and ASCT in pediatric solid tumor. However, there is no randomized clinical study to evaluate the efficacy of prophylactic use of anti-fungal agent to date.

Itraconazole is one of newly developed antifungal agents and many physicians started to use itraconazole as first-line antifungal agent in the management of neutropenic fever in immunocompromised patients. However, the efficacy of prophylactic itraconazole has not been established in children with solid tumor, especially who receive HDCT and ASCT.

In this context, we are going to evaluate the efficacy of prophylactic use of itraconazole in children with high-risk solid tumors during HDCT and ASCT. "Prophylactic" group will be treated with itraconazole once ANC fall below 500/uL regardless of infection and "Empirical" group will be treated with itraconazole only when high fever persists despite of treatment with first-line anti-bacterial agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high risk solid tumors who are going to receive high dose chemotherapy and autologous hematopoietic stem cell transplantation

Exclusion Criteria:

* Significant organ toxicity (National Cancer Institute [NCI] grade > 2) prior to high dose chemotherapy and autologous hematopoietic stem cell transplantation

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-06 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Presence/absence of documented fungal infection | until post transplant day 30
Presence/absence of clinical fungal infection | until post transplant day 30
Total duration of high fever | until post transplant day 30
Total duration of antibiotic treatment | until post transplant day 30

CONTACTS AND LOCATIONS:
Overall Officials: KiWoong Sung, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim YJ, Sung KW, Hwang HS, Jung SH, Kim JY, Cho EJ, Lim SJ, Choi YB, Cheuh HW, Lee SH, Yoo KH, Koo HH. Efficacy of itraconazole prophylaxis for autologous stem cell transplantation in children with high-risk solid tumors: a prospective double-blind randomized study. Yonsei Med J. 2011 Mar;52(2):293-300. doi: 10.3349/ymj.2011.52.2.293. PMID 21319349